CLINICAL TRIAL: NCT00125541
Title: Pharmacokinetics, Clinical Efficacy and Safety of C1 Inhibitor Concentrate (C1-Esteraseremmer-N) for the Treatment of Hereditary (and Acquired) Angioedema
Brief Title: C1-Esteraseremmer-N for the Treatment of Hereditary (and Acquired) Angioedema
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Responsible Party: P. Strengers, Sanquin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KB2003.01C
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Angioedema
Keywords: MeSH: angioneurotic edema, complement 1 inactivators; Hereditary Angioedema Type I or II, Acquired Angioedema
MeSH Terms: conditions — Angioedema; Hereditary Angioedema Types I and II; Acquired angioedema

INTERVENTIONS:
Drug: C1 inhibitor concentrate (C1-esteraseremmer-N) — every 5-7 days

SUMMARY:
A multicentre study to investigate the pharmacokinetics, clinical efficacy and safety of nanofiltered Cetor® (called C1-esteraseremmer-N during the development phase) for the treatment of hereditary angioedema (HAE) will be performed. This study (KB2003.01) consists of three parts: Part A - pharmacokinetics (phase II); Part B - treatment of attacks of angioedema (phase III); and Part C - prophylactic use of C1 inhibitor (phase III). Parts B + C will provide data on the efficacy of C1-esteraseremmer-N.

The changes within the manufacturing process of C1-esteraseremmer-N, compared to Cetor® nanofiltration and omission of hepatitis B immunoglobulin, most likely will not affect tolerability. The nanofiltration will provide more safety regarding viruses.

In part C of the study, a number of HAE patients will be treated prophylactically with open-label C1-esteraseremmer-N for a period of 16 weeks. The number of attacks occurring will be compared with historical data. If possible, also some patients treated prophylactically with C1 inhibitor for acquired angioedema will be included.

DETAILED DESCRIPTION:
A multicentre study to investigate the pharmacokinetics, clinical efficacy and safety of nanofiltered Cetor® (called C1-esteraseremmer-N during the development phase) for the treatment of hereditary angioedema (HAE) will be performed. This study (KB2003.01) consists of three parts: Part A - pharmacokinetics (phase II); Part B - treatment of attacks of angioedema (phase III); and Part C - prophylactic use of C1 inhibitor (phase III). Parts B + C will provide data on the efficacy of C1-esteraseremmer-N.

The changes within the manufacturing process of C1-esteraseremmer-N, compared to Cetor® nanofiltration and omission of hepatitis B immunoglobulin, most likely will not affect tolerability. The nanofiltration will provide more safety regarding viruses.

In part C of the study, a number of HAE patients will be treated prophylactically with open-label C1-esteraseremmer-N for a period of 16 weeks. The number of attacks occurring will be compared with historical data. If possible, also some patients treated prophylactically with C1 inhibitor for acquired angioedema will be included.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for hereditary angioedema patients:

* Established diagnosis of hereditary angioedema type I or II: markedly decreased C1 inhibitor activity; decreased (type I), normal or elevated (type II) level of C1 inhibitor antigen; decreased level of C4.
* Patients already using C1 inhibitor concentrate for prophylaxis of angioedema attacks.
* Age ≥ 16 years
* Signed informed consent by patient and patient's legal representative if under 18 years old

Inclusion criteria for acquired angioedema patients:

* Established diagnosis of acquired angioedema: recurrent attacks of angioedema without urticaria; no family history; decreased functional C1 inhibitor; decreased level of C4.
* Autoantibodies to C1 inhibitor or decreased C1q or onset after the third decade of life.
* Age ≥ 16 years
* Patient already using C1 inhibitor concentrate for prophylaxis of angioedema attacks
* Signed informed consent by patient and patient's legal representative if under 18 years old

Exclusion Criteria:

Exclusion criteria for hereditary angioedema patients:

* Use of angioedema prophylactic medication during the study, other than C1-esteraseremmer-N.
* Change in oral contraceptives starting from the last two months before the start of the trial until the end of the study period.
* Presence of clinically relevant C1 inhibitor auto antibodies
* Participation in another pharmaceutical clinical study, which can interfere with this study, in the last 3 months prior to the study, other than in part A of this protocol.
* Usage of heparin starting from the last two days prior to the study until the end of the study period.
* B-cell malignancy
* Pregnancy or lactation
* History of allergic reaction to C1 inhibitor concentrate or other blood products

Exclusion criteria for acquired angioedema patients:

* Participation in another pharmaceutical clinical study, which can interfere with this study, in the last 3 months prior to the study
* Usage of heparin within the last two days prior to the study
* Pregnancy or lactation
* History of allergic reaction to C1 inhibitor concentrate or other blood products

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary objective in this clinical study is to evaluate the prevention of angioedema attacks in patients prophylactically treated with C1-esteraseremmer-N. | 16 weeks

SECONDARY OUTCOMES:
The secondary objective of this study is to evaluate the safety and clinical activity of C1-esteraseremmer-N. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: M. M. Levi, Prof. Dr., Principal Investigator — Academic Medical Centre Amsterdam
Locations (1):
- Academic Medical Centre, Amsterdam, Netherlands